CLINICAL TRIAL: NCT00312507
Title: Surfactant Lavage vs. Bolus Surfactant in Neonates With Meconium Aspiration
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1000007730
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2006-10

CONDITIONS: Meconium Aspiration Syndrome
Keywords: Meconium Aspiration Syndrome; Surfactant; Bronchoalveolar Lavage; newborns
MeSH Terms: conditions — Meconium Aspiration Syndrome

INTERVENTIONS:
Drug: Bovine Lipid Extract Surfactant (administered by lavage)
Drug: Bovine Lipid Extract Surfactant (administered by bolus)

SUMMARY:
The objective of this pilot study is to examine the feasibility and safety of performing a larger trial to assess outcomes following treatment of meconium aspiration syndrome with surfactant lavage compared to bolus surfactant. Specifically, we will determine if surfactant lavage results in a more rapid improvement in physiologic outcomes (e.g. pulmonary compliance), as well as clinical outcomes (e.g. length of time on mechanical ventilation).

DETAILED DESCRIPTION:
Meconium-stained amniotic fluid occurs in about 5 to 20% of all births in the United States, with meconium aspiration syndrome occuring in approximately 5% of these infants. In this disease process, meconium is believed to mechanically obstruct the airways, causing a chemical pneumonitis and inactivate surfactant. Approximately one-third of these babies need mechanical ventilation and approximately 5% die. Since 1990 surfactant has been the standard of care for treatment of respiratory distress syndrome. Pulmonary compliance and gas exchange often improve rapidly after administration of surfactant. Its use has led to significantly reduced mortality rates and improved short-term respiratory function. There is evidence to support its use in other neonatal respiratory disorders where there is dysfunction or inactivation of surfactant. Its use in meconium aspiration syndrome is the most well-studied alternate use to date. The Canadian Pediatric Society's (2005) position statement recommends that infants with meconium aspiration syndrome who are intubated and require more than 50% oxygen should receive exogenous surfactant therapy.

Studies in both animals and humans suggest that surfactant helps in meconium aspiration, either administered as a bolus or as a lavage. There have been no trials to date comparing the efficacy of surfactant lavage to bolus surfactant in human neonates with meconium aspiration or examining the physiologic effects of surfactant, given as either a bolus or lavage, in the treatment of meconium aspiration syndrome. This study will assess the relative efficacy of these two methods of administering surfactant and their effect on physiologic and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* infants ≥ 36 weeks gestational age with evidence of meconium aspiration syndrome
* respiratory support (ventilator or CPAP) within 6 h of birth
* enrolment within 24 h of birth
* significant difficulty with oxygenation, as indicated by an oxygenation index (OI) > 15, where OI = (FiO2 x MAP) / PaO2 and MAP is the mean airway pressure
* presence of an arterial line

Exclusion Criteria:

* major congenital anomalies
* known antenatal diagnosis of significant congenital heart disease (diagnosis other than patent foramen ovale, patent ductus arteriosus or small ventricular septal defect)
* infants with a maternal history of oligohydramnios and physical features consistent with the diagnosis
* surfactant administration prior to enrolment
* hemodynamic instability defined as intractable hypotension on more than 2 inotropes
* significant pulmonary hemorrhage, defined as pulmonary hemorrhage in association with a 30% (absolute) increase in FiO2 and radiologic changes consistent with pulmonary hemorrhage
* significant intracranial hemorrhage, defined as a unilateral or bilateral Grade III or IV intraventricular hemorrhage or a large intracranial, non-intraventricular hemorrhage
* significant illness meeting ECMO criteria with an OI > 40
* infants in whom withdrawal of intensive care is likely

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20
Dates: Start 2006-04

PRIMARY OUTCOMES:
% change in oxygenation indices from baseline to 1 and 6 h following treatment
% change in dynamic pulmonary compliance from baseline to 1 and 6 h following treatment
% change in pulmonary artery pressure from baseline to 1 and 6 h following treatment
measures of efficacy of ventilation and oxygenation at 1 h and 6 h following treatment
cardiac function by echocardiography at 6 hours following treatment

SECONDARY OUTCOMES:
% change in oxygenation indices, dynamic pulmonary compliance and pulmonary vascular resistance from baseline to 12, 24 and 48 h following treatment
measures of efficiency of ventilation and oxygenation at 12, 24 and 48 h following treatment
duration of mechanical ventilation, defined as the cumulative time of mechanical ventilation
length of time on CPAP
length of time with oxygen supplementation
length of time on inotropes and maximum inotropic score.
need for and length of use of NO
need for and length of use of ECMO
time to full enteral feeds
attainment of exit criteria
development of significant pulmonary hemorrhage
development of significant intracranial hemorrhage
development of tension pneumothorax requiring drainage
need for repeat surfactant
length of stay in a level III NICU
mortality

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McNamara, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada